CLINICAL TRIAL: NCT03150576
Title: Randomised, Phase II/III, 3 Stage Trial to Evaluate the Safety and Efficacy of the Addition of Olaparib to Platinum-based Neoadjuvant Chemotherapy in Breast Cancer Patients With TNBC and/or gBRCA.
Brief Title: Platinum and Polyadenosine 5'Diphosphoribose Polymerisation Inhibitor for Neoadjuvant Treatment of Triple Negative Breast Cancer and/or Germline BRCA Positive Breast Cancer
Acronym: PARTNER
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK (Other)
Responsible Party: Principal Investigator, Prof. Jean Abraham, Professor, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PARTNER
Record Dates: First submitted 2016-07-26; First posted 2017-05-12 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Triple negative breast cancer; germline BRCA; platinum and PARP inhibitor; neoadjuvant chemotherapy; olaparib
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — olaparib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): 4 cycles of: Paclitaxel 80mg/m2 Day 1, 8 & 15, every 3 weeks, Carboplatin area under the curve (AUC) 5 Day 1, every 3 weeks
  Interventions: Drug: Paclitaxel and Carboplatin
- Research 1 (Experimental): 4 cycles of: Paclitaxel 80mg/m2 on Days 1, 8 & 15 every 3 weeks, Carboplatin AUC 5 Day 1, every 3 weeks, Olaparib oral 150mg twice daily, Day -2 to Day 10 every 3 weeks
  Interventions: Drug: Olaparib; Drug: Paclitaxel and Carboplatin
- Research 2 (Experimental): 4 cycles of: Paclitaxel 80mg/m2 on Days 1, 8 & 15 every 3 weeks, Carboplatin AUC 5 Day 1, every 3 weeks, Olaparib oral 150mg twice daily, Day 3 to Day 14 every 3 weeks
  Interventions: Drug: Olaparib; Drug: Paclitaxel and Carboplatin

INTERVENTIONS:
Drug: Olaparib — Patients will self-administer Olaparib by mouth. Olaparib tablets should be taken twice daily at the same time each day approximately 12 hours apart.
  Other Names: Lynparza
  Arms: Research 1; Research 2
Drug: Paclitaxel and Carboplatin — Paclitaxel I.V. 80mg/m2 in 0.9% sodium chloride 500ml or according to local practice, will be given over 60 minutes on days 1, 8 & 15, every 3 weeks for 4 cycles. Carboplatin I.V. AUC5 in 5% dextrose 500ml or according to local practice, over 30-60minutes on day 1 every 3 weeks for 4 cycles.
  Other Names: Taxol and Paraplatin

SUMMARY:
This neoadjuvant trial for patients with TNBC and/or gBRCA breast cancer, aims to investigate the safety and efficacy (improvement in pathological Complete Response at surgery) of concurrent platinum-based chemotherapy with olaparib an inhibitor of the PARP enzyme (PARPi).

DETAILED DESCRIPTION:
Randomised, phase II/III 3 stage trial to evaluate the safety and efficacy of the addition of olaparib to platinum-based neoadjuvant chemotherapy in breast cancer patients with TNBC and/or gBRCA.

Disease under investigation: Breast Cancer

Purpose of clinical trial: To establish if the addition of olaparib to neoadjuvant platinum-based chemotherapy for Triple Negative Breast Cancer (TNBC) and/or germline BRCA (gBRCA) breast cancer is safe and improves efficacy.

Trial Design: Open label, randomised, 3-stage Phase II/III

Sample Size: Minimum of 780 patients (including at least 220 gBRCA patients equally allocated to the control and the selected research arm).

Non Investigational Medicinal Products: Prophylactic granulocyte-colony stimulating factor (G-CSF) to be given as per local practice and 3 cycles of anthracyclines as per local practice.

Treatment period: A minimum of 21 weeks of chemotherapy followed by surgery.

Procedures: Screening & enrolment

Eligible patients with early breast cancer will be registered and consented for screening:

BRCA mutation test Tumour Infiltrating Lymphocytes(TILs) score Cytokeratin 5/6 (CK5/6), Epidermal Growth Factor Receptor (EGFR) +/-, Androgen Receptor (AR) status by Immunohistochemistry (IHC).

Standard assessment prior to chemotherapy Standard staging to exclude metastatic disease. When eligibility is confirmed, patients will be randomised via a web-based central system which will allocate each patient a unique randomisation number associated with one of the treatment arms.

PARTNERing Pathway - For those patients who still have residual disease after receiving neoadjuvant chemotherapy +/- olaparib there is the opportunity to be screened to a sub-study to receive a further two cycles of chemotherapy consisting of Duralumab and AZD6738.

End of Trial: For patients, the end of trial is after the last follow-up visit or contact with the research team planned 10 years after surgery.

Procedures for safety monitoring during trial: Pharmacovigilance will be performed by the PARTNER Trial Office. Also, the Trial Management Group and the Independent Data and Safety Monitoring Committee will regularly review the patient safety data.

Criteria for discontinuation of trial treatment on safety grounds:

Severe toxicity or inter-current illness, requiring cessation in the judgement of patient's clinician.

Patient within 4 weeks has not recovered from toxicity to an extent that allows further treatment.

Patient unable to comply with trial procedures. Disease progression while on trial treatment. Patient becomes pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 and 70.
* Written informed consent, willing and able to comply with the Protocol for the duration of the trial including undergoing treatment and scheduled visits and examinations.
* Histologically confirmed invasive breast cancer.
* ER-negative*, and HER2-negative** breast cancer (TNBC). Patients will be eligible with any PR status but PR expression must be scored.

OR

* Germline BRCA (gBRCA) mutation positive, HER2 negative, and PgR / ER of any status.
* T1, T2 or T3 tumours.
* T4 tumour of any size with direct extension to (a) chest wall or (b) skin. OR Inflammatory carcinoma with tumour of any size. OR

Other Locally Advanced Disease:

* Involvement of ipsilateral large or fixed axillary lymph nodes, or infra or supraclavicular nodes (>10mm diameter or clinical N2 or N3) and primary breast tumour of any diameter.
* Involvement of ipsilateral large or fixed axillary lymph nodes, or infra or supraclavicular nodes (>10mm diameter, or clinical N2 or N3), without a primary breast tumour identified, the presence of breast cancer in a Lymph Node (LN) must be histopathologically confirmed by LN biopsy.

OR

Multifocal tumour:

- with at least one tumour with a size>10mm.

* Patients with bilateral disease are eligible to enter the trial provided that both breast disease meets the above criteria.
* Be fit to receive the trial chemotherapy regimen in the opinion of the responsible clinician:

Adequate bone marrow, hepatic, and renal function. ECOG performance status of 0, or 1.

* Treatment should be commenced within 6 weeks of the diagnostic biopsy. In uncommon circumstances, where medically acceptable, treatment is permitted to start within a maximum of 9 weeks of the diagnostic biopsy.
* Availability of the Tumour Infiltrating Lymphocytes score is required.
* Availability of CK 5/6 and EGFR +/- Androgen Receptor IHC score.
* Availability of slides and paraffin embedded tissue blocks from pre-chemotherapy core biopsy and from primary surgical resection is required.
* Women of child-bearing potential (WCBP), defined as not surgically sterilized or not post-menopausal for at least 24 consecutive months if age ≤55 year or 12 months if age >55 years, must have a negative serum or urine pregnancy test within 14 days prior to randomisation.
* All WCBP and all sexually active male patients as well as their partners must be aware that they should not conceive during the treatment period and therefore should routinely use effective forms of contraception, throughout their participation in the trial and for at least 6 months after the last dose of trial treatment. Please follow the olaparib contraception guidelines.

Exclusion Criteria:

* T0 tumour in absence of axillary node >10mm.
* TNBC with a non-basal phenotype which strongly expresses Androgen Receptor.
* Previous or concomitant chemotherapy or biological agents used for the treatment of cancer in the last 5 years.
* Malignancy within the last 5 years except: adequately treated non-melanoma skin cancer; curatively treated in situ cancer of the cervix; ductal carcinoma in situ (DCIS); Stage 1, grade 1 endometrial carcinoma; or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia.
* Evidence of distant metastasis apparent prior to randomisation.
* Patients with uncontrolled seizures.
* Pre-existing sensory or motor neuropathy of CTCAE v4.03, grade ≥2.
* Concomitant use of known potent CYP3A4 inhibitors and inducers. Consider wash-out periods.
* Pregnant or breast feeding women.
* Not suitable for neoadjuvant chemotherapy in the opinion of the responsible clinician.
* Major surgery within 14 days of starting trial treatment and patients must have recovered from any effects of any major surgery.
* Any evidence of other disease or any concomitant medical or psychiatric problems which in the opinion of the Investigator would prevent completion of treatment or follow-up. For example:

Evidence of severe or uncontrolled cardiac disease Uncontrolled ventricular arrhythmia Recent myocardial infarction (within 12 months) Active infection including Hepatitis B, Hepatitis C and Human Immunodeficiency virus (HIV). Screening for chronic conditions is not required.

* ECG with mean resting QTc >470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the trial medication
* Known hypersensitivity to olaparib, carboplatin, paclitaxel or their excipients (including cremophor).
* Whole blood transfusions in the last 120 days prior to blood sampling for BRCA test as it may interfere with the results (packed red blood cells and platelet transfusions are acceptable).

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2016-05; Primary Completion 2024-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Stage 1 - Number of participants with treatment-related adverse events as assessed by NCI CTCAE v4.03. | 1 year - when first 25 patients in each research arm who had received at least one dose of Olaparib protocol treatment have completed their protocol treatment.
  Primary outcome measure - safety of the addition of olaparib to three weekly carboplatin/weekly paclitaxel chemotherapy.
Stage 2 - pCR rate and completion rate of Olaparib treatment as per protocol. | 15 months - when pathological complete response (pCR) is available for 53 patients in each of two research arms.
  Primary outcome measure - pCR in each of the two research arms. At the end of stage 2, one of the research treatments will be dropped using the 'pick the winner' method.
Stage 3 - Efficacy analysis based on pCR at surgery. To be assessed by central review of pathology reports. | 5.5 years - October 2021 approx.
  Primary outcome measure - pCR at surgery after neoadjuvant treatment. pCR rates after neoadjuvant chemotherapy +/- olaparib, defined as no residual invasive carcinoma within the breast (Ductal Carcinoma in situ permitted) AND no evidence of metastatic disease within the lymph nodes.

SECONDARY OUTCOMES:
pCR at surgery - assessed by review of histopathology slides | Up to 2 years after last patient randomised
  pCR at surgery assessed by central pathology review of the diagnosis and surgery slides.
PARTNERing Pathway | 2 cycles (each lasting 28 days)
  For those patients who still have residual disease after receiving neoadjuvant chemotherapy there is the opportunity to receive a further two cycles of Duralumab and AZD6738. Durvalumab I.V will be administered on cycle 1, day 1 and cycle 2, day 1. AZD6738 will be self administered by patients by mouth twice a day for 7 days beginning on cycle 1, day 22 and cycle 2, day 22.
Relapse-Free Survival (RFS) | Up to 10 years after last patient is randomised
  Relapse Free Survival (RFS), calculated from date of randomisation to date of first relapse or date of death from all causes, whichever occurs first.
Breast cancer specific survival (BCSS) | Up to 10 years after last patient is randomised
  Breast cancer specific survival (BCSS), calculated from date of randomisation to date of death from breast cancer.
Distant disease-free survival | Up to 10 years after last patient is randomised
  Distant disease-free survival, calculated from date of randomisation to date of the first distant disease relapse or date of death from all causes, whichever occurs first.
Local recurrence-free survival | Up to 10 years after last patient is randomised
  Local recurrence-free survival, calculated from date of randomisation to date of the first local recurrence or date of death from all causes, whichever occurs first.
Overall survival (OS) | Up to 10 years after last patient is randomised
  Overall survival (OS), calculated from date of randomisation to date of death from all causes.
Time to second cancer (TTSC) | Up to 10 years after last patient is randomised
  Time to second cancer (TTSC), calculated from the date of randomisation to the date of diagnosis of second cancer.
pCR in breast alone | Up to 2 years after last patient is randomised
  pCR in breast alone
Residual Cancer Burden (RCB) | Up to 10 years after last patient is randomised
  Residual Cancer Burden (RCB) I-III will be assessed by central pathology review.
Radiological response - as assessed by radiological response criteria as per RECIST v1.1 | Up to 2 years after last patient is randomised
  Radiological response after 4th and final cycles
Treatment related toxicities - as assessed by CTCAE v4.03 | Up to 10 years after last patient is randomised
  Treatment related toxicities
Quality of Life Questionnaire | Up to 10 years after last patient is randomised
  Quality of Life (sub-study). Questionnaire to be completed by patient prior to start of treatment, following cycle 4 and cycle 7, following surgery and then annually for two years to document long-term effects on quality of life.

OTHER OUTCOMES:
Discovery and validation of markers that can be correlated with outcomes (pCR and RFS). | Up to 15 years after last patient is randomised
  Discovery and validation of prognostic, pharmacogenetic and pharmacogenomic markers that can be correlated with outcomes (pCR and RFS) in patients randomised to received olaparib compared with those who are not.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Abraham, Principal Investigator — The University of Cambridge, Department of Oncology
Locations (30):
- United Kingdom (30):
  - Cambridge University Hospitals NHS Foundation Trust & the University of Cambridge, Cambridge, Cambridgeshire
  - Queen's Hospital, Burton-on-Trent, Derby
  - The Christie, Manchester, Lancs
  - Pinderfields General Hospital, Wakefield, Yorkshire
  - University Hospital Ayr, Ayr
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Bedford General Hospital, Bedford
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Haematology & Cancer Centre, Bristol
  - West Suffolk Hospital, Bury St Edmunds
  - Velindre Cancer Centre, Cardiff
  - Colchester General Hospital, Colchester
  - Russells Hall Hospital, Dudley
  - Hinchingbrooke Hospital, Huntingdon
  - Ipswich Hospital, Ipswich
  - Kidderminster General Hospital, Kidderminster
  - University Hospital Crosshouse, Kilmarnock
  - University College London Hospital, London
  - Royal Free Hospital, London
  - Mount Vernon Cancer Centre, Northwood
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Peterborough City Hospital, Peterborough
  - Poole Hospital, Poole
  - The Alexandra Hopsital, Redditch
  - Queen's Hospital, Romford
  - Southampton General Hospital, Southampton
  - Singleton Hospital, Swansea
  - Royal Hampshire County Hospital, Winchester
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: Yes
All Clinical Trial data will be considered to be shared on formal application to the Trial CI & TMG, however data affecting or considered as having the potential to affect the integrity or the endpoints of the trial and/or other collaborations will not be shared (or until such time that they no longer are deemed to have an effect).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: While the trial is on-going: dependant on specific request. After the end of the trial: (as per our funding T&Cs) data will be released into an open-source web repository.
Access Criteria: Formal application to the Partner TMG and Chief Investigator.

REFERENCES:
- [Derived] Abraham JE, O'Connor LO, Grybowicz L, Alba KP, Dayimu A, Demiris N, Harvey C, Drewett LM, Lucey R, Fulton A, Roberts AN, Worley JR, Chhabra MA, Qian W, Brown J, Hardy R, Vallier AL, Chan S, Cidon MEU, Sherwin E, Chakrabarti A, Sadler C, Barnes J, Persic M, Smith S, Raj S, Borley A, Braybrooke JP, Staples E, Scott LC, Palmer CA, Moody M, Churn MJ, Pilger D, Zagnoli-Vieira G, Wijnhoven PWG, Mukesh MB, Roylance RR, Schouten PC, Levitt NC, McAdam K, Armstrong AC, Copson ER, McMurtry E, Galbraith S, Tischkowitz M, Provenzano E, O'Connor MJ, Earl HM; PARTNER Trial Group. Neoadjuvant PARP inhibitor scheduling in BRCA1 and BRCA2 related breast cancer: PARTNER, a randomized phase II/III trial. Nat Commun. 2025 May 13;16(1):4269. doi: 10.1038/s41467-025-59151-0. PMID 40360463
- [Derived] Abraham JE, Pinilla K, Dayimu A, Grybowicz L, Demiris N, Harvey C, Drewett LM, Lucey R, Fulton A, Roberts AN, Worley JR, Chhabra A, Qian W, Vallier AL, Hardy RM, Chan S, Hickish T, Tripathi D, Venkitaraman R, Persic M, Aslam S, Glassman D, Raj S, Borley A, Braybrooke JP, Sutherland S, Staples E, Scott LC, Davies M, Palmer CA, Moody M, Churn MJ, Newby JC, Mukesh MB, Chakrabarti A, Roylance RR, Schouten PC, Levitt NC, McAdam K, Armstrong AC, Copson ER, McMurtry E, Tischkowitz M, Provenzano E, Earl HM. The PARTNER trial of neoadjuvant olaparib with chemotherapy in triple-negative breast cancer. Nature. 2024 May;629(8014):1142-1148. doi: 10.1038/s41586-024-07384-2. Epub 2024 Apr 8. PMID 38588696
- [Derived] Woitek R, McLean MA, Ursprung S, Rueda OM, Manzano Garcia R, Locke MJ, Beer L, Baxter G, Rundo L, Provenzano E, Kaggie J, Patterson A, Frary A, Field-Rayner J, Papalouka V, Kane J, Benjamin AJV, Gill AB, Priest AN, Lewis DY, Russell R, Grimmer A, White B, Latimer-Bowman B, Patterson I, Schiller A, Carmo B, Slough R, Lanz T, Wason J, Schulte RF, Chin SF, Graves MJ, Gilbert FJ, Abraham JE, Caldas C, Brindle KM, Sala E, Gallagher FA. Hyperpolarized Carbon-13 MRI for Early Response Assessment of Neoadjuvant Chemotherapy in Breast Cancer Patients. Cancer Res. 2021 Dec 1;81(23):6004-6017. doi: 10.1158/0008-5472.CAN-21-1499. Epub 2021 Oct 8. PMID 34625424